CLINICAL TRIAL: NCT02554292
Title: Post MArket Surveillance of SeQuent Please Neo With ScORing Balloon Lesion Preparation in Real WorlD Patients
Brief Title: Post Market Surveillance of SeQuent Please Neo With Scoring Balloon
Acronym: PASSWORD
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: Ernst von Bergmann Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AAG-O-A-1507
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Drug Coated Balloon Angioplasty, Scoring Balloon Dilatation — Percutaneous Coronary Intervention
  Other Names: SeQuent® Please Neo Drug Coated Balloon, NSE Alpha Scoring Balloon

SUMMARY:
The main objective of the SeQuent® Please Neo post market surveillance is to assess the clinical suitability of the combination of pre-dilatation using the NSE Alpha scoring balloon before the use of the paclitaxel-coated SeQuent® Please Neo in an 'all comer'/ 'real world' setting for the treatment of in-stent restenosis and de-novo lesions.

DETAILED DESCRIPTION:
The aim of this post market surveillance is to document the safety and efficacy of the drug-coated balloon Sequent® Please Neo in combination with the NSE Alpha scoring balloon in the treatment of both in-stent restenosis and de-novo lesions in native coronary arteries with reference diameters of 2.5 mm up to 4.0 mm with lesion lengths of 30 mm for procedural success and preservation of vessel patency

ELIGIBILITY:
Inclusion Criteria:

* patients with in-stent restenosis and de-novo lesions in coronary arteries

Exclusion Criteria:

* Intolerance to paclitaxel and/or the balloon coating
* Allergy to components of the balloon coating
* Pregnancy and lactation
* Complete occlusion of the treatment vessel
* Severely calcified stenosis
* Cardiogenic shock
* Risk of an intraluminal thrombus
* Haemorrhagic diathesis or another disorder such as gastro-intestinal ulceration or cerebral circulatory disorders which restrict the use of platelet aggregation inhibitor therapy and anti-coagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease, specifically with in-stent restenosis
Sampling Method: Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure | 9 months
  Target Vessel Failure = TLR + Myocardial Infarction (MI) + cardiac death

SECONDARY OUTCOMES:
procedural success rate | intraprocedural
  lesion crossing success in in-stent restenotic lesions
Target Lesion Revascularization rate = Re-PCI + CABG(TLR) | 9 months
cardiac death | 9 months
  death of cardiac or unknown causes
Rate of coronary arterial bypass grafting (CABG) | 9 months
rate of myocardial infarction | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bonaventura, MD, Principal Investigator — Klinikum Ernst von Bergmann
Locations (1):
- Klinikum Ernst von Bergmann, Potsdam, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wohrle J, Zadura M, Mobius-Winkler S, Leschke M, Opitz C, Ahmed W, Barragan P, Simon JP, Cassel G, Scheller B. SeQuentPlease World Wide Registry: clinical results of SeQuent please paclitaxel-coated balloon angioplasty in a large-scale, prospective registry study. J Am Coll Cardiol. 2012 Oct 30;60(18):1733-8. doi: 10.1016/j.jacc.2012.07.040. Epub 2012 Oct 3. PMID 23040575
- [Background] Almalla M, Schroder JW, Pross V, Stegemann E, Marx N, Hoffmann R. Everolimus-eluting versus paclitaxel-eluting stents for treatment of bare metal stent restenosis. Am J Cardiol. 2011 Aug 15;108(4):518-22. doi: 10.1016/j.amjcard.2011.03.080. Epub 2011 May 31. PMID 21624553
- [Result] Kufner S, Cassese S, Valeskini M, Neumann FJ, Schulz-Schupke S, Hoppmann P, Fusaro M, Schunkert H, Laugwitz KL, Kastrati A, Byrne RA; ISAR-DESIRE 3 Investigators. Long-Term Efficacy and Safety of Paclitaxel-Eluting Balloon for the Treatment of Drug-Eluting Stent Restenosis: 3-Year Results of a Randomized Controlled Trial. JACC Cardiovasc Interv. 2015 Jun;8(7):877-84. doi: 10.1016/j.jcin.2015.01.031. Epub 2015 May 20. PMID 26003022
- [Result] Rittger H, Brachmann J, Sinha AM, Waliszewski M, Ohlow M, Brugger A, Thiele H, Birkemeyer R, Kurowski V, Breithardt OA, Schmidt M, Zimmermann S, Lonke S, von Cranach M, Nguyen TV, Daniel WG, Wohrle J. A randomized, multicenter, single-blinded trial comparing paclitaxel-coated balloon angioplasty with plain balloon angioplasty in drug-eluting stent restenosis: the PEPCAD-DES study. J Am Coll Cardiol. 2012 Apr 10;59(15):1377-82. doi: 10.1016/j.jacc.2012.01.015. Epub 2012 Feb 29. PMID 22386286
- [Result] Byrne RA, Neumann FJ, Mehilli J, Pinieck S, Wolff B, Tiroch K, Schulz S, Fusaro M, Ott I, Ibrahim T, Hausleiter J, Valina C, Pache J, Laugwitz KL, Massberg S, Kastrati A; ISAR-DESIRE 3 investigators. Paclitaxel-eluting balloons, paclitaxel-eluting stents, and balloon angioplasty in patients with restenosis after implantation of a drug-eluting stent (ISAR-DESIRE 3): a randomised, open-label trial. Lancet. 2013 Feb 9;381(9865):461-7. doi: 10.1016/S0140-6736(12)61964-3. Epub 2012 Dec 1. PMID 23206837
- [Result] Xu B, Gao R, Wang J, Yang Y, Chen S, Liu B, Chen F, Li Z, Han Y, Fu G, Zhao Y, Ge J; PEPCAD China ISR Trial Investigators. A prospective, multicenter, randomized trial of paclitaxel-coated balloon versus paclitaxel-eluting stent for the treatment of drug-eluting stent in-stent restenosis: results from the PEPCAD China ISR trial. JACC Cardiovasc Interv. 2014 Feb;7(2):204-211. doi: 10.1016/j.jcin.2013.08.011. PMID 24556098
- [Derived] Bonaventura K, Schwefer M, Yusof AKM, Waliszewski M, Krackhardt F, Steen P, Ocaranza R, Zuhdi AS, Bang LH, Graf K, Bock U, Chin K. Systematic Scoring Balloon Lesion Preparation for Drug-Coated Balloon Angioplasty in Clinical Routine: Results of the PASSWORD Observational Study. Adv Ther. 2020 May;37(5):2210-2223. doi: 10.1007/s12325-020-01320-2. Epub 2020 Apr 9. PMID 32274746